CLINICAL TRIAL: NCT06403865
Title: Evaluation en Vie réelle de la qualité de Vie de Personnes Vivant Avec le VIH traité Par cabotégravir et Rilpivirine Par Patient-Reported Outcomes
Brief Title: Patient-Reported Outcomes in Real-life of Cabotegravir and Rilpivirine
Acronym: PANTER
Status: Not yet recruiting | Type: Observational
Sponsor: University Paris 7 - Denis Diderot (Other)
Collaborators: Hopital Foch (Other)
Responsible Party: Principal Investigator, Dr Martin Duracinsky, PhD, MD, Assistance Publique - Hôpitaux de Paris
Other Study IDs: PANTER Quanti
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Quality of Life
Keywords: Long-Acting Injectable Regimen; HIV; Patient-reported Outcomes; Treatment switch
MeSH Terms: interventions — cabotegravir, rilpivirine drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PLWHIV: People living with HIV-1
  Interventions: Drug: Cabotegravir, Rilpivirine Drug Combination

INTERVENTIONS:
Drug: Cabotegravir, Rilpivirine Drug Combination — Treatment switch to CAB+RPV LA

SUMMARY:
Context The introduction of the long-acting injectable antiretroviral treatment cabotegravir and rilpivirine into the therapeutic armamentarium for people living with HIV represents a potentially significant evolution in patients' experience of their treatment and pathology. Its effects on the quality of life of PLHIV are explored in this research. In addition, the two-monthly intra-muscular injection regimen also raises questions about the city-to-hospital transition of care for PLHIV, as well as compliance with the therapeutic window.

Main objective To evaluate the effect of switching HIV treatment to CAB+RPV LA on health-related quality of life on the "Treatment Impact" dimension of the PROQOL-HIV questionnaire, 15 months after switching treatment.

Population People living with HIV-1 whose ARV treatment has been changed to an injectable CAB+RPV LA treatment

Study Design Observational study. Inclusion at HIV medical follow-up visit for change of ARV treatment to CAB/RPV.

Self-administered questionnaires at M3, M9 and M15 after change of treatment (first CAB/RPV injection).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 carriers
* Patients who changed treatment (as part of routine care) to injectable CAB+RPV at the same visit as the inclusion visit
* HIV-RNA less than or equal to 50 copies/mL for at least 6 months prior to inclusion visit
* Patient 18 years of age or older
* Patient able to read, understand and answer self-questionnaires in French

Exclusion Criteria:

* Pregnant or breast-feeding women
* Known hypersensitivity to cabotegravir or rilpivirine
* Documented resistance to cabotegravir or rilpivirine
* Chronically active hepatitis B (HBsAg+)
* Any pathology or history of treatment which, in the investigator's judgment, would contraindicate the patient's inclusion in the study or prevent him/her from following the constraints of the protocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People living with HIV-1 whose ARV treatment has been changed to an injectable CAB+RPV LA treatment
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Treatment Impact - PROQOL-HIV | between D0 (baseline) and 15 months after the first injection of CAB+RPV LA
  Evolution of the score of the "Treatment impact (TI)" dimension of the PROQOL-HIV questionnaire (10 items)

IPD SHARING:
Plan to Share IPD: No